CLINICAL TRIAL: NCT03014739
Title: Evaluation of the Reproducibility of Young's Modulus and Shear Wave Velocity Measurements With SWE™ in Achilles Tendons and Plantar Fascia
Brief Title: Evaluation of Shear Wave Elastography Reproducibility in Achilles Tendons and Plantar Fascia
Acronym: ME1
Status: Completed | Type: Observational
Sponsor: SuperSonic Imagine (Industry)
Collaborators: Beijing Chao Yang Hospital (Other); Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ME1
Record Dates: First submitted 2016-12-14; First posted 2017-01-09 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Achilles Tendon; Plantar Fascia
Keywords: Elastography; Musculoskeletal System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Supersonic ShearWave Elastography — ShearWave Elastography (SWE) is part of routine ultrasound examination

SUMMARY:
Achilles tendon plays a significant role in walking and sporting activities, particularly through ankle joint and lower limbs stability. Ultrasound imaging can be the first-line examination of choice for patients suspected of having Achilles tendon injury, which is more and more frequent. Nowadays, ultrasound elastography can be used to evaluate the viscoelasticity properties of Achilles tendon, however little is known about the reproducibility of the technique. This study aims to evaluate the reproducibility of supersonic shear imaging SWE™ Young's modulus measurements of shear wave velocity (m/s) in Achilles tendon and plantar fascia.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with normal Achilles tendon:
* Normal adult aged over 18 years old;
* Without lower limb malformation;
* With no symptoms of Achilles tendon lesion and no negative results of routine ultrasound examination for a possible tendinopathy.

Exclusion Criteria:

* Subjects who failed to meet all inclusion criteria were will be automatically excluded;
* Subjects who did will not wish or could will not sign the informed consent in person.
* Volunteers with abnormal Achilles tendon for any of these reasons:

  * Lower limb malformation;
  * Achilles tendon pain, Achilles tendon disease, surgical history of Achilles tendon surgery, morphologic abnormalities of Achilles tendon ( gray-scale/color Doppler/MRI/plain film);
  * Suffer from systemic, metabolic and endocrine diseases, including but not limited to, diabetes, familial hyperlipidemia (FH), systemic lupus erythematosus (SLE), gout, ankylosing spondylitis, hyperthyroidism, chronic renal failure, etc.
  * Pregnant women;
  * Apply Ongoing hormone hormonal therapy;
  * Athletes

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers without any Achilles tendon disease
Sampling Method: Non-Probability Sample
Enrollment: 1165 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Intra- and inter-operator reproducibility | Baseline
  Intraclass Correlation Coefficient

OTHER OUTCOMES:
Effect of limb dominance | Baseline
  Variability of ICC as a function of dominant versus non-dominant leg

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Chao-Yang Hospital, Beijing
  - The third Affiliated Hospital of Peking University, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cao W, Sun Y, Liu L, Wang Z, Wu JY, Qiu L, Wang YX, Yuan Y, Shen SF, Chen Q, Chen T, Zhang W, Wu CJ, Liu FX, Zhong SG, Chen L, Tong MH, Cui LG, Guo RJ. A Multicenter Large-Sample Shear Wave Ultrasound Elastographic Study of the Achilles Tendon in Chinese Adults. J Ultrasound Med. 2019 May;38(5):1191-1200. doi: 10.1002/jum.14797. Epub 2018 Sep 12. PMID 30208234